CLINICAL TRIAL: NCT01584869
Title: Emergency Capsule Endoscopy in Severe GI-bleeding
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23042012
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: GI-bleeding
Keywords: GI-bleeding; capsule endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capsule endoscopy (Experimental)
  Interventions: Device: capsule endoscopy

INTERVENTIONS:
Device: capsule endoscopy

SUMMARY:
Primary objective: Evaluation of capsule endoscopy in the emergency setting of severe GI-Bleeding.

ELIGIBILITY:
Inclusion Criteria:

patients with signs of severe GI-bleeding (with melena or dark bloody stool) and hemodynamic instability (defined as (pre)collapse or MAP < 80 mmHg or HR > 110) and/or drop of hemoglobin > 2g/dl/d and/or need of transfusion of minimum of 2 packed red cells

Exclusion Criteria:

missing consent form, pregnancy, origin of bleeding found in upper GI-endoscopy (e.g. blood in the stomach, ulcer, varices with signs of bleeding, mallory-weiss-tear, Angiodysplasia (with signs of bleeding), refluxesophagitis LA C or D) fresh bloody stool, known stenosis of the bowel, known site of bleeding, known inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the influence of capsule endoscopy on guidance of further diagnostic or therapeutic procedures. | after complete recruitment

SECONDARY OUTCOMES:
frequency of mid-GI-bleeding in all patients
diagnostic yield | after complete recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, München, Bavaria, Germany

REFERENCES:
- [Derived] Schlag C, Menzel C, Nennstiel S, Neu B, Phillip V, Schuster T, Schmid RM, von Delius S. Emergency video capsule endoscopy in patients with acute severe GI bleeding and negative upper endoscopy results. Gastrointest Endosc. 2015 Apr;81(4):889-95. doi: 10.1016/j.gie.2014.09.035. PMID 25432532